CLINICAL TRIAL: NCT01636869
Title: Plasma Concentrations of Bupivacaine After Spinal Anesthesia With Single Shot Femoral Nerve Block and Peri-articular Injection in Total Knee Arthroplasty
Brief Title: Plasma Concentrations of Bupivacaine After Peri-articular Injection in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Saowaphak Lapmahapaisan, instructor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 010/2555
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Serum Bupivacaine Level; Periarticular Block; Total Knee Arthroplasty
Keywords: bupivacaine level; periarticular block; total knee arthroplasty
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bupicavaine (Experimental)
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — 20 ml of 0.5% bupivacaine for single-shot femoral nerve block will be done at the beginning then another 20 ml of 0.5% bupivacaine for periarticular block will be performed at the end of operation.
  Blood sample will be drawn at 60 min after femoral nerve block and before periarticular block, 15, 30, 45, 60 min after periarticular block.

SUMMARY:
Patients with knee arthroplasty usually performed under spinal anesthesia with a single-shot femoral nerve block and periarticular block, so we would like to know the plasma concentration of bupivacaine in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age of 30-70 yr
* ASA I-II
* patient undergo total knee arthroplasty under spinal block and single shot femoral nerve block and periarticular block

Exclusion Criteria:

* patient's refusal
* allergic to bupivacaine
* body weight less than 50 kg
* liver disease
* heart disease
* coagulopathy
* Hct<35%
* infection at both groin

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
plasma concentration of bupivacaine after spinal anesthesia with single-shot femoral nerve block and periarticular block | 2 hours

SECONDARY OUTCOMES:
bupivacaine toxicity | 24 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand